CLINICAL TRIAL: NCT03377608
Title: Modifiers of Tenofovir Exposure in the Female Genital Tract of African Women on Depo-provera
Brief Title: Modifiers of Tenofovir in the Female Genital Tract
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: MU-JHU CARE (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000171
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: HIV/AIDS; Contraception
Keywords: tenofovir; microbiome; inflammation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Inflammation | interventions — Tenofovir; Medroxyprogesterone Acetate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Depo-Provera
  Interventions: Drug: Tenofovir Disoproxil Fumarate; Drug: Depo-Provera
- Non-hormonal contraception
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Two cervical biopsies, blood plasma, PBMC, urine, and two cervicovaginal swabs will be collected at a single study visit
Drug: Depo-Provera — Two cervical biopsies, blood plasma, PBMC, urine, and two cervicovaginal swabs will be collected at a single study visit
  Groups: Depo-Provera

SUMMARY:
Two-armed, single visit, pharmacokinetic study to compare tenofovir diphosphate concentrations in cervical tissues of women on Depo-Provera contraception vs non-hormonal contraception.

ELIGIBILITY:
Inclusion Criteria:

* Female, or transgender female with a cervix, aged 18-35 years old
* HIV-positive
* Stable on antiretroviral regimen containing TDF for at least 2 weeks at time of enrollment.
* Virally suppressed (HIV-RNA copies <50 copies/mL) for at least 6 months at time of enrollment.
* Willing to refrain from vaginal intercourse and use of vaginal devices such as douches and sex toys within 72 hours of the biopsy visit.
* Willing and able to give signed informed consent.

Exclusion Criteria:

* Currently pregnant or previous pregnancy within 3 months of enrollment
* Currently breast feeding
* Symptomatic vaginal infection within 2 weeks prior to enrollment
* Unexplained, undiagnosed abnormal bleeding per vagina, bleeding per vagina during or following vaginal intercourse, or gynecologic surgery within 90 days prior to enrollment
* History of vulvar/vaginal/ cervical dysplasia, neoplasia or cancer, atypical squamous cells of undetermined significance, condyloma, or human papilloma virus (HPV) in the past year
* Use of oral and/or vaginal preparations of antibiotic or antifungal medications within 30 days prior to the enrollment visit

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women will be recruited from an existing cohort.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Cervical Tissue Concentrations | Day 1
  Assess the influence of hormonal contraception on tenofovir concentrations in cervical tissues

SECONDARY OUTCOMES:
Proinflammatory cytokines | Day 1
  To determine relationship between local inflammation and drug disposition in the female genital tract
Gene expression of drug metabolizing enzymes and transporters | Day 1
  To assess the influence of hormonal contraception on the expression of drug metabolizing enzymes and transporters in cervical tissue
Vaginal microbiome | Day 1
  To identify potential role of the vaginal microbiome in local drug disposition

CONTACTS AND LOCATIONS:
Locations (1):
- MU-JHU Care Ltd, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicol MR, Eneh P, Nakalega R, Kaiser T, Kabwigu S, Isingel E, Beksinska M, Sykes C, Fowler MG, Brown TT, Staley C, Kiweewa Matovu F. Depot Medroxyprogesterone Acetate and the Vaginal Microbiome as Modifiers of Tenofovir Diphosphate and Lamivudine Triphosphate Concentrations in the Female Genital Tract of Ugandan Women: Implications for Tenofovir Disoproxil Fumarate/Lamivudine in Preexposure Prophylaxis. Clin Infect Dis. 2020 Apr 10;70(8):1717-1724. doi: 10.1093/cid/ciz443. PMID 31131846